CLINICAL TRIAL: NCT00476931
Title: A Phase 2 Repeat Dosing Clinical Trial of SB-509 in Subjects With Moderate to Severe Diabetic Neuropathy and Unmeasurable Nerve Conduction Velocity
Brief Title: Clinical Trial of SB-509 in Subjects With Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SB-509-0701
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Polyneuropathy
Keywords: Diabetic neuropathy; Diabetes Type 1 or 2; Moderate to severe sensorimotor diabetic polyneuropathy; Unmeasurable nerve conduction velocity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SB-509
  Interventions: Biological: SB-509
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SB-509 — 60 mg dose
  Arms: 1
Other: Placebo — Saline
  Arms: 2

SUMMARY:
The purpose of the study is to study the clinical effects of the investigational drug, SB-509 versus placebo in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
SB-509 contains the gene (DNA-a kind of biological "blueprint") for a protein. When a researcher injects SB-509 into your legs, the drug enters the muscle and nerve cells around the injection site and causes these cells to make a protein. This protein causes your cells to increase production of another protein called vascular endothelial growth factor (VEGF), which may improve the structure and function of nerves. In addition, there are changes in the levels of 28 additional proteins in your cells. These proteins function to promote the growth of cells, are structures in cells, help synthesize products, and affect immune cells, and some have unknown functions. This increase in your own VEGF proteins may protect and repair the damaged nerves caused by diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

* Have a clinical diagnosis of diabetes mellitus type I or II for at least 12 months prior to the study.
* Have received a diagnosis of moderate to severe sensorimotor diabetic neuropathy from a neurologist (a doctor who specializes in disorders of the nervous system) or endocrinologist (a doctor who specializes in diabetes). This type of neuropathy is a loss of sensation and muscle function that occurs in the legs and hands in a stocking and glove distribution. Subjects with diabetic neuropathy that results in loss of sensation or muscle function in only one nerve and results in loss of nerve function of the blood vessels and causes low blood pressure, will not be eligible.
* Unmeasurable nerve conduction velocity in any lower extremity nerve: peroneal, tibial or sural due to diabetic polyneuropathy
* If female and of childbearing potential, agree to use a medically acceptable physical barrier method during the study.
* Have blood pressure < 140/90 mm Hg
* Body mass index (BMI) < 38 kg/m2

Key Exclusion Criteria:

Subjects with the following are NOT eligible to participate in this study:

* Have moderate to severe ischemic heart disease, any history of congestive heart failure, or have had a myocardial infarction (heart attack) within the previous 6 months.
* Have chronic foot or leg ulcers for >1 month, gangrene in the legs, or any previous amputation of the lower extremity.
* Have a history of cancer within the past 5 years (except for curable non-melanoma cancer of the skin, superficial bladder cancer in complete remission, or any other cancer that has been in complete remission for at least 5 years).
* Have colon polyps. If patients have a history of benign colonic polyps that have been removed, they must have evidence of a normal colonoscopy within the last 12 months.
* Require any drug that depresses patients' immune systems (such as methotrexate, cyclophosphamide, or cyclosporine) when they receive the study drug and for 30 days afterwards.
* Have a known disorder that affects patients' immune systems (such as HIV/AIDS, hepatitis B virus [HBV], hepatitis C virus [HCV], sarcoidosis, tuberculosis, rheumatoid arthritis, or autoimmune disorders).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Total Neuropathy Score (TNS),Evoked nerve conduction velocity (NCV), Quantitative Sensory Testing (QST), %of subjects with conversion of unmeasurable to measurable NCV and NIS-LL | One year

SECONDARY OUTCOMES:
Safety | One year

CONTACTS AND LOCATIONS:
Locations (20):
- United States (19):
  - Coordinated Clinical Research, La Jolla, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Torrance Clinical Research, Lomita, California
  - SF Clinical Research Center, San Francisco, California
  - Diablo Clinical Research, Walnut Creek, California
  - Bradenton Research Center, Bradenton, Florida
  - Neurology Clinical Research, Sunrise, Florida
  - Laszlo J. Mate', M.D., West Palm Beach, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Creighton Diabetes Center, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Upstate Clinical Research, Albany, New York
  - Peripheral Neuropathy Center, Weill Medical College of Cornell University, New York, New York
  - Neurological Institute Columbia University College of Physicians and Surgeons, New York, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Diabetes Center of the Southwest, Midland, Texas
  - DGD Research, San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Instituto Mexicano de Investigación Clinica, Mexico City, Col. Roma, Mexico

REFERENCES:
- See also: Related Info — http://www.sangamo.com